CLINICAL TRIAL: NCT01987115
Title: Comparison of Fascial Manipulation With Traditional Physiotherapy for the Treatment of Trigger Fingers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorin Daniel Iordache (Other)
Responsible Party: Sponsor-Investigator, Sorin Daniel Iordache, Head of Hand Surgery, Beilinson Hospital, Clalit Health Services
Organization: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMTF-1
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Trigger Finger
Keywords: Trigger Finger; Physiotherapy; Fascial Manipulation
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fascial Manipulation (Experimental): Group will receive fascial manipulation at 3 centers of coordination (C.C) at: 1. C.C above the pronator teres muscle. (M.F unit of INTRA-CUBITUS), 2. C.C above proximal part of pronator quadratus muscle, between the palmaris longus and the flexor carpi radialis tendons (M.F unit of INTRA-CARPUS), 3. C.C in the mid-palmar region between metacarpus 3-4 (M.F unit of INTRA-DIGIT).4. C.C. over the muscle belly of Ext. Digit and Ext. Pollicis Longus (M.F unit of EXTRA-CARPUS).
  Interventions: Procedure: Fascial manipulation
- Traditional physiotherapy (Active Comparator): Group will receive U.S. treatment delivered to the A1 pulley area (3 Megahertz, over 1cm², for 5 minutes), Metacarpophalangeal and Proximal interphalangeal joint mobilization (for 5 minutes), eccentric stretching, and self exercises at home (self-stretch and self-massage).
  Interventions: Procedure: Traditional physiotherapy

INTERVENTIONS:
Procedure: Fascial manipulation — Group will receive fascial manipulation at 3 centers of coordination (C.C) at: 1. C.C above the pronator teres muscle. (M.F unit of INTRA-CUBITUS), 2. C.C above proximal part of pronator quadratus muscle, between the palmaris longus and the flexor carpi radialis tendons (M.F unit of INTRA-CARPUS), 3. C.C in the mid-palmar region between metacarpus 3-4 (M.F unit of INTRA-DIGIT).4. C.C. over the muscle belly of Ext. Digit and Ext. Pollicis Longus (M.F unit of EXTRA-CARPUS).
  Arms: Fascial Manipulation
Procedure: Traditional physiotherapy — Group will receive U.S. treatment delivered to the A1 pulley area (3 Megahertz, over 1cm², for 5 minutes), Metacarpophalangeal and Proximal interphalangeal joint mobilization (for 5 minutes), eccentric stretching, and self exercises at home (self-stretch and self-massage).
  Arms: Traditional physiotherapy

SUMMARY:
Trigger finger is a relatively common disorder affecting the hand. There is limited evidence on the efficiency of traditional physiotherapy in treating this condition. Fascial manipulation is a gaining momentum manual therapy method. To our knowledge the efficiency of fascial manipulation techniques in the treatment of trigger finger was not reported. The purpose of this study is to investigate the efficiency of the technique and to compare it with the traditional physiotherapy treatment.

DETAILED DESCRIPTION:
All adult patients diagnosed with a trigger finger by the primary investigator will be eligible for the study. Criteria for diagnosing the condition are a history of catching of the involved finger accompanied by pain over the A1 pulley on the volar aspect of the hand. Exclusion criteria include patients with a locked finger (SST Grade IV on the Quinell classification as modified by Green (18)), age younger than 18, traumatic trigger fingers (post-surgery or fracture in the distal forearm or hand), patient with low pain tolerance (hyperalgesia/allodynia etc.), trigger thumbs, multiple (more than 1) and recurrent trigger fingers or patients who received additional treatments for this finger in the past year, motor vehicle or work accidents or patients with additional compensation claims, patients with conditions that may cause secondary catching including tumors involving the finger or the joint, inflammatory conditions especially rheumatoid arthritis, and patients with osteoarthritis involving the specific metacarpo-phalangeal joint. Patients who cannot commit to attend the planned therapeutic sessions will also be excluded from the study.

All the subjects will be informed of the study and consented will be obtained. The patients will be randomized in two groups based on drawing a closed envelope from a box containing an equal number of notes for the respective therapeutic protocols. Each patient will undergo 8 sessions of therapy over a period of 6 weeks.

Group A protocol includes U.S. treatment delivered to the A1 pulley area (3 MHz, over 1cm², for 5 minutes), MP and PIP joint mobilization (for 5 minutes), eccentric stretching, and self exercises at home (self-stretch and self-massage).

Group B protocol will receive fascial manipulation including deep kneading of muscular fascia at 3 centers of coordination (C.C) at: 1. C.C above the pronator teres muscle. (M.F unit of INTRA-CUBITUS), 2. C.C above proximal part of pronator quadratus muscle, between the palmaris longus and the flexor carpi radialis tendons (M.F unit of INTRA-CARPUS), 3. C.C in the mid-palmar region between metacarpus 3-4 (M.F unit of INTRA-DIGIT).

Demographic data including the age and gender, and previous medical history will be recorded. The duration of the symptoms and the fingers involved will be noted. The patients will undergo a brief assessment including the determination of the SST according to the modified Quinell classification, and the determination of the number of triggering events occurring in 10 active flexion/extension cycles. The grip power (average of 3 times) and pinch will be measured using dynamometers. An x-ray of the involved hand will be obtained to rule out concomitant conditions in the hand. The patients will be asked to fill a Quick Dash questionnaire and a VAS chart.

A similar assessment will be repeated at 6 weeks by an independent assessor, who will be blinded to the protocol which was used.

Six months from the end of the treatment a mail survey will be conducted in patients in whom the treatment succeeded. The survey will include information about recurrence of the condition (No recurrence, occasional pain or catching, or full recurrence) a VAS scale and the Quick DASH questionnaire.

We consider a difference of 1.5 points in VAS between the two treatment groups at 6 weeks to be clinically significant. Assuming a 20% decrease in VAS with traditional physiotherapy, considering an α value of 0.05 and a β value of 0.2 to obtain 80% statistical power, and allowing for a 35% lost to follow-up, we plan to recruit 70 patients for this study, 35 patients in each treatment group.

The data will be recorded and the statistical analysis will be performed using the Microsoft Excel Spreadsheet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with trigger finger by primary investigator
* Adult
* Good command of Hebrew

Exclusion Criteria:

* Locked finger
* Younger than 18
* Secondary triggers (Post-traumatic, tumor, rheumatic disease, pregnancy, etc.)
* Low pain tolerance (hyperalgesia/allodynia etc.)
* Trigger thumbs
* Multiple trigger fingers
* Recurrent trigger finger
* Patient received additional treatments
* Patients with compensation claims
* Patients who cannot commit to attend the planned therapeutic sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-11; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for pain | 6 weeks
  Decrease in pain as measured by a visual analog scale at 6 weeks

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand score | 6 weeks
  Decrease in the The Disabilities of the Arm, Shoulder and Hand at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sorin D Iordache, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Migdal Hamea Clinic Clalit Health Services, Tel Aviv, Israel